CLINICAL TRIAL: NCT05435846
Title: A Multicenter Phase I/Ib Study of Capmatinib Plus Trametinib in Patients With Metastatic MET Exon 14 Skipping Mutation Positive NSCLC
Brief Title: Capmatinib Plus Trametinib for the Treatment of Metastatic Non-small Cell Lung Cancer With MET Exon 14 Skipping Mutation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Collin Blakely (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Collin Blakely, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22653; NCI-2022-04800 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer
Keywords: MET exon 14 skipping mutation; Mutation Positive
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — capmatinib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1: Dose Escalation (Experimental): Patients receive 200 - 400 mg capmatinib orally, twice a day and 1.0 or 1.5 mg trametinib orally once a day on days 1-28 of each cycle. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capmatinib; Drug: Trametinib
- Phase 1b: Dose Expansion (Experimental): Patients will receive the recommended phase 2 dose (RP2D) or capmatinib in combination with trametinib determined by the safety profile of the Phase 1 group. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Capmatinib; Drug: Trametinib

INTERVENTIONS:
Drug: Capmatinib — Given orally
  Other Names: INC280
Drug: Trametinib — Given orally
  Other Names: TMT212; Mekinist

SUMMARY:
This phase I/Ib trial studies the side effects and best doses of capmatinib plus trametinib when given together for the treatment of patients with MET exon 14 skipping mutation non-small cell lung cancer that has spread to other places in the body (metastatic). Capmatinib is in a class of medications called kinase inhibitors. It works by blocking the action of an abnormal protein that signals cancer cells to multiply. This helps slow or stop the spread of cancer cells. Trametinib is in a class of medications called kinase inhibitors. It works by blocking the action of an abnormal protein that signals cancer cells to multiply. This helps stop the spread of cancer cells. Capmatinib and trametinib are "targeted therapies." These targeted therapies work by detecting and targeting a mutation in the MET gene. Giving Capmatinib and trametinib may kill more tumor cells in patients with metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify recommended phase II dose (RP2D) of capmatinib in combination with trametinib in non-small cell lung cancer (NSCLC) with MET 14 exon mutation, MET amplification, or MET fusion (Phase I).

II. To further characterize the safety profile of the RP2D of capmatinib in combination with trametinib in MET-exon14 mutated NSCLC (Phase Ib).

SECONDARY OBJECTIVES:

I. To further characterize the safety profile of the combination of capmatinib and trametinib in NSCLC with MET exon 14 mutation, MET amplification, or MET fusion (Phase I).

II. To determine preliminary efficacy ofcapmatinib in combination with trametinib in MET-exon14 mutated NSCLC (Phase Ib)

EXPLORATORY OBJECTIVES:

I. To evaluate the pharmacokinetics of capmatinib in combination with trametinib.

II. To identify biomarkers of response to capmatinib and trametinib. III. To identify mechanisms of resistance tocapmatinib and trametinib.

OUTLINE: This is a phase I dose-escalation study of capmatinib and trametinib followed by a phase Ib dose expansion study.

Patients receive capmatinib orally (PO) twice daily (BID) and trametinib PO once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 12 months

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed, non-small cell lung cancer.
* Documented MET exon 14 skipping mutation by tumor DNA sequencing or cell-free DNA assay by Clinical Laboratory Improvement Act (CLIA) - approved laboratory AND previously received treatment with a MET inhibitor (capmatinib crizotinib, savolitinib, or tepotinib) with evidence of disease progression, in the opinion of the investigator.

  * Note - MET inhibitor therapy is NOT required to be the most recent anti-cancer therapy. Prior treatment with platinum-based chemotherapy or anti-programmed cell death protein 1 (PD-1) /programmed death-ligand 1 (PD-L1) therapy (alone or in combination with chemotherapy) is allowed, but not required.
* - or (For dose escalation only): MET amplification or fusion detected in tumor sample or cell-free DNA by next generation sequencing (NGS) or Fluorescent in situ hybridisation (FISH) by CLIA-approved laboratory AND prior treatment with a MET inhibitor (capmatinib crizotinib, savolitinib, or tepotinib) with at least 5 months of clinical benefit, followed by disease progression, in the opinion of the investigator.
* Archived tissue available or willingness to undergo new tumor biopsy.
* Measurable disease defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
* Life expectancy of at least 3 months.
* Age >= 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 (Karnofsky) > 60%.
* Resolution of all acute toxic effects (other than alopecia, or non-clinically significant lab abnormalities) of prior chemotherapy, targeted therapy, immunotherapy, radiotherapy, or surgical procedures to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 grade 1.
* Absolute neutrophil count >= 1,500/microliter (mcL)
* Platelets >= 100,000/mcL
* Hemoglobin (Hgb) >= 9 g/dl
* Total bilirubin within 1.2 X institutional upper limit of normal, unless elevated due to Gilbert's syndrome and direct bilirubin is within normal limits.
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT)) =< 3 X institutional upper limit of normal if no known liver metastases.
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase (SGPT)) =< 3 X institutional upper limit of normal if no known liver metastases.
* Alkaline phosphatase (ALP) =< 5.0 X institutional upper limit of normal.
* Creatinine =< 1.5 x within institutional upper limit of normal.

  * Creatinine glomerular filtration rate (GFR) >= 30 mL/min/1.73 m^2,calculated using the Cockcroft-Gault equation, unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m^2.
* Asymptomatic serum amylase =< grade 2.

  * Asymptomatic serum amylase increase grade 1 and 2 are allowed if at the beginning of the study is confirmed to have no signs and/or symptoms suggesting pancreatitis or pancreatic injury (e.g., elevated P-amylase, abnormal imaging findings of pancreas, etc.)
* Serum lipase =< upper limits of normal (ULN).
* Ability to understand a written informed consent document, and the willingness to sign it.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Individuals with a history of hepatitis C virus (HCV) infection must have been treated and cured or currently be on treatment with an undetectable HCV viral load.
* Individuals with treated brain metastases are eligible if follow-up brain imaging (within 1 month prior to first dose) after central nervous system (CNS)-directed therapy shows no evidence of progression and not on steroids.
* Individuals with a prior or concurrent malignancy are eligible for this trial as long as they are not on active treatment and no active disease is present, and whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen. Exceptions: thyroid hormone replacement is allowed and adjuvant hormonal therapy for breast cancer is allowed.
* Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 16 weeks after last administration of study treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 16 weeks after last administration of study treatment.

Exclusion Criteria:

* Known activating mutations or oncogenic fusions in Epithelial Growth Factor Receptor (EGFR), KRAS g12c, ALK, ROS1, Neurotrophic tyrosine receptor kinase (NTRK), BRAF V600E, or RET or known on-target MET mutations on residues D1228 or Y1230.
* For Phase I patients enrolling into dose levels 1 or -1, intolerability of prior treatment with capmatinib 300 mg BID requiring dose reduction or permanent discontinuation is exclusionary.
* For Phase I patients enrolling into dose level -2, intolerability of prior treatment with capmatinib 200 mg BID requiring dose reduction or permanent discontinuation is exclusionary.
* For Phase I patients enrolling into dose level 2, intolerability of prior treatment with capmatinib 400 mg BID requiring dose reduction or permanent discontinuation is exclusionary.
* Phase Ib patients enrolling into the dose expansion cohort must have previously tolerated the RP2D of capmatinib if they have received prior capmatinib treatment.
* Pregnant women are excluded from this study because capmatinib and trametinib are tyrosine kinase inhibitors (TKIs) with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with capmatinib and trametinib, breastfeeding should be discontinued if the mother is treated with capmatinib and trametinib.
* Patients who have received systemic anti-cancer therapies within the following time periods prior to the first dose of study drug: within 3 weeks of cytotoxic chemotherapy or antibody therapy, radiation within 2 weeks, targeted therapy within 7 days.

  * Note: Concomitant administration of Luteinizing hormone-releasing hormone (LHRH) analogues for prostate cancer and somatostatin analogues for neuroendocrine tumors are allowed as per standard of care. Patients who are currently receiving and progressing on capmatinib monotherapy will be allowed to continue treatment without interruption
* History of interstitial lung disease or pneumonitis.

  * Note: History of radiation pneumonitis not requiring steroids is allowed.
* Known Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) infection, or human immunodeficiency virus (HIV) with inadequate CD4+ T cell counts or a history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections.

  * Note: Participants with laboratory evidence of cleared HBV and HCV infection will be permitted). Patients living with HIV, with adequate CD4+ T cell counts, and without a history of AIDS-defining opportunistic infections will be permitted.
* Known active COVID-19 infection.

  * Note: Patients who have recovered from an infection and test negative for viral ribonucleic acid (RNA) will be allowed.
* History or evidence of cardiovascular risk including any of the following:

  * Left ventricular ejection fraction (LVEF) < lower limit of normal (LLN) by echocardiogram (ECHO) or multigated acquisition scan (MUGA).
  * A QT interval corrected for heart rate using the Fridericia's formula (QTcF) 470 msec.
  * History or evidence of current clinically significant uncontrolled arrhythmias.
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to study enrollment.
  * History or evidence of current >= Class II congestive heart failure as defined by New York Heart Association (NYHA).
  * Treatment refractory hypertension defined as a blood pressure of systolic > 150 mmHg and/or diastolic > 95 mm Hg which cannot be controlled by anti-hypertensive therapy.
* Patients with intra-cardiac defibrillators.

  * Note: Participants with atrial fibrillation controlled (defined as not requiring change in cardiac drug dosing, emergency room visit, or hospital admission) for >30 days prior to dosing are eligible.
* Is currently receiving any other investigational agents.
* Hypersensitivity to capmatinib or trametinib or any of its excipients.
* Patients with known history or current evidence of retinal vein occlusion (RVO) or retinal pigment epithelial detachment (RPED).
* Major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) within 4 weeks prior (2 weeks for resection of brain metastases) to starting study treatment or who have not recovered from side effects of such procedure.

  * Note: Video-assisted thoracic surgery (VATS) and mediastinoscopy will not be counted as major surgery and participants can be enrolled in the study >= 1 week after the procedure.
* Participants receiving treatment with strong inducers of CYP3A that cannot be discontinued at least 1 week prior to the start of treatment with study treatment and for the duration of the study.
* Any condition that in the opinion of the investigator would interfere with the participant's safety or compliance while on trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with reported dose limiting toxicity (DLT) (Phase I) | 1 cycle (each cycle is 28 days)
  Proportion of participants who experience a DLT for capmatinib in combination with trametinib in Phase I. A dose limiting toxicity (DLT) will be defined as any adverse event that are considered by the investigator to be at least possibly related to capmatinib or trametinib and are observed during the first 28 days of treatment (Cycle 1).
Proportion of participants with treatment-emergent adverse events (Phase Ib) | Up to 12 months
  Proportion of participants with treatment-emergent Adverse Events, will be reported as preferred terms using Medical Dictionary for Regulatory Activities (MedDRA).as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 5.0) in Phase Ib (Dose Expansion).

SECONDARY OUTCOMES:
Proportion of participants with treatment-emergent adverse events (Phase I) | From initiation of study treatment until 30 days post-treatment discontinuation
  Proportion of participants with Adverse Events, as graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 5.0 in Phase Ib
Overall Response Rate (ORR) (Phase Ib) | Up to 12 months
  The ORR is defined as the best overall response recorded from the start of the treatment until disease progression or recurrence assessed over a 1-year period from the start of treatment using RECIST version 1.1 criteria. The percentages of patients with a best overall response rate of complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) will be determined.
Mean Disease Control Rate (DCR) (Phase Ib) | Up to 12 months
  DCR will be defined as the percentage of patients who have achieved CR, PR, or SD (based on RECIST 1.1 criteria) for at least 12 weeks. The mean DCR and the standard deviation of DCR will be summarized.
Median Progression Free Survival (PFS) (Phase Ib) | Up to 12 months
  PFS will be calculated as 1+ the number of days from the first dose of study drugs to documented radiographic progression or death due to any cause. For patients who continue treatment post-progression, the date of radiographic progression will be used for PFS analysis. The Kaplan-Meier analysis will be used to calculate the median PFS with 95% confidence interval.
Overall survival (OS) (Phase Ib) | Up to 12 months
  OS will be calculated as 1+ the number of days from the first dose of study drugs to death due to any cause. The Kaplan-Meier analysis will be used to calculate the median PFS with 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Collin M Blakely, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No